CLINICAL TRIAL: NCT05248685
Title: Single-center, Open-Label, Non-randomized, Single-Arm Phase 1 Study to Evaluate the Safety and Tolerability of Optimized Dual CD33/CLL1 CAR T Cells in Subjects With Refractory or Relapsed Acute Myeloid Leukemia
Brief Title: Optimized Dual CD33/CLL1 CAR T Cells in Subjects With Refractory or Relapsed Acute Myeloid Leukemia
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: no patients
Sponsor: Beijing Boren Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BRYY-IIT-LCYJ-2021-026
Record Dates: First submitted 2022-01-17; First posted 2022-02-21 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Acute Myeloid Leukemia
Keywords: CAR-T; Leukemia; Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Leukemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Dual CD33/CLL1 CAR T (Experimental): All patients who receive Dual CD33/CLL1 CAR T Cell infusion
  Interventions: Biological: Dual CD33/CLL1 CAR T

INTERVENTIONS:
Biological: Dual CD33/CLL1 CAR T — Subjects will be pretreated with chemotherapy prior to infusion of CAR T cells: After the collection of PBMC and about 5 days before infusion, lymphodepletion chemotherapy (fludarabine at 30 mg/m^2/day and cyclophosphamide at 250 mg/m^2/day) will be administrated for 3 days. Then this study will be using BOIN1/2 approach from starting dose 1: 1×10^6 (±20%) to dose 2: 5×10^6 (±20%). If the manufactured cells were not sufficient to meet the preassigned standard dose criteria, patients are given infusion at a low dose of 5×10^5 (±20%)

SUMMARY:
This is a single-center, open-label, non-randomized, single-arm Phase 1 Study to evaluate safety and tolerability of optimized Dual CD33/CLL1 CAR T Cells in subjects with refractory or relapsed acute myeloid leukemia. Maximum of twenty subjects will be enrolled. After the collection of PBMC and about 5 days before infusion, lymphodepletion chemotherapy (fludarabine at 30 mg/m^2/day and cyclophosphamide at 250 mg/m^2/day) will be administrated for 3 days.

Then this study will be using BOIN1/2 approach from starting dose 1: 1×10^6 (±20%) to dose 2: 5×10^6 (±20%). If the manufactured cells were not sufficient to meet the preassigned standard dose criteria, patients are given infusion at a low dose of 5×10^5 (±20%) /kg.

ELIGIBILITY:
Inclusion Criteria:

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

1. Co-expression of tumor surface antigens CD33 and CLL1 was confirmed (among which, the proportion of cells expressing CD33 was ≥ 80%; and the proportion of cells expressing CLL1 ≥ 80%); patients with primary drug resistance, chemotherapy relapse, extramedullary relapse, persistent residual disease positive or relapsed/refractory acute myeloid leukemia after allogeneic hematopoietic stem cell transplantation;
2. Male or female, aged 1-70 years;
3. No serious allergic constitution;
4. Eastern Cooperative Oncology Group (ECOG) performance status (Oken et al., 1982) score 0 to 2;
5. Have life expectancy of at least 60 days based on investigator's judgement;
6. Provide a signed informed consent before any screening procedure; subjects who voluntarily participate in the study should have the ability to understand and sign the informed consent form and be willing to follow the study visit schedule and relevant study procedure, as specified in the protocol. Candidates aged 19-70 years need to be sufficiently conscious and able to sign the treatment consent form and voluntary consent form; Children candidates of 8-18 years old need to be sufficiently conscious and able to sign the treatment consent form and voluntary consent form and their legal guardian or patient advocate has also need to sign the treatment consent form and voluntary consent form, respectively.Children candidates of 1-7 can be recruited after the legal guardian or patient advocate has signed the treatment consent form and voluntary consent form.

Exclusion Criteria:

An individual who meets any of the following criteria will be excluded from participation in this study:

1. Intracranial hypertension or disorder of consciousness;
2. Symptomatic heart failure or severe arrhythmia;
3. Symptoms of severe respiratory failure;
4. Complicated with other types of malignant tumors;
5. Diffuse intravascular coagulation;
6. Serum creatinine and / or blood urea nitrogen ≥ 1.5 times of the normal value;
7. Suffering from septicemia or other uncontrollable infections;
8. Patients with uncontrollable diabetes;
9. Severe mental disorders;
10. Obvious and active intracranial lesions were detected by cranial magnetic resonance imaging (MRI);
11. Have received organ transplantation (excluding bone marrow transplant);
12. Reproductive-aged female patients with positive blood HCG test;
13. Screened to be positive of infection of hepatitis (including hepatitis B and C), AIDS or syphilis;
14. For patients with CAR-T cells derived from autologous lymphocytes, leukemia blasts accounted for more than 30% of all cells in peripheral blood;
15. Patients unable to provide a transplant donor about 30 days after the CAR-T cell transfusion.

Ages: 1 Year to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-02-16 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Dose limiting toxicity (DLT) | 21 days post intravenous injection
  DLT assessment according to the clinical study protocol
Incidence and severity of adverse events (AE) | 30 days post intravenous injection

SECONDARY OUTCOMES:
Objective response rate (ORR) | 28 days post infusion
  Objective response rate (ORR) according to NCCN, Complete response (CR),CR with incomplete blood count recovery (CRi)
Concentration of PK CAR positive T cells in peripheral blood | 30 days post infusion
  Proliferation and survival of CAR T cells in peripheral blood.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Boren Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided